CLINICAL TRIAL: NCT06297005
Title: The Impact of E-cigarettes During Pregnancy on Childhood Health Outcomes (ECHO) Study.
Brief Title: The Impact of E-cigarettes During Pregnancy on Childhood Health Outcomes Study
Acronym: ECHO
Status: Recruiting | Type: Observational
Sponsor: University College Dublin (Other)
Collaborators: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: 21/FFP-P/10154
Record Dates: First submitted 2024-02-16; First posted 2024-03-06 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Vaping; Pregnancy Related; Pediatric Respiratory Diseases
Keywords: Vaping; Pregnancy; Paediatric health
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine for cotinine measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vapers: Women who vape during pregnancy
- Smokers: Women who smoke tobacco during pregnancy
- Controls: Women who neither smoke tobacco or vape during pregnany

SUMMARY:
Tobacco smoking in pregnancy is now widely accepted as having adverse health outcomes for both the mother and fetus. Tobacco smoking in pregnancy is associated with increased incidence of miscarriage, stillbirth and preterm birth as well as low birthweight, respiratory infections, wheeze and asthma in childhood. E-cigarettes are a popular method for trying to quit smoking in Ireland and there has been an explosion in the use of e-cigarettes over the past ten years. However, there is currently insufficient evidence on their long-term safety and effectiveness as a smoking cessation tool. E-cigarettes contain varying combinations of compounds and flavours which are used differently in different e-cigarette types, with unknown long-term effects. Research has shown that pregnant women perceive e-cigarettes to be a healthier option when compared with tobacco smoking. But, there is very little known about the long-term health impact of exposure of unborn babies to e-cigarettes during pregnancy.

The ECHO study will determine what the long-term health outcomes are in children born to mothers who use e-cigarettes during pregnancy. Specifically, we will focus on birth, nutritional, brain development and respiratory outcomes in children. To answer this research question, the ECHO study will recruit infants born to women who use e-cigarettes during pregnancy across three maternity hospitals and follow them up over 2 years. We will invite women at their booking visit to take part in this research study. We plan to also recruit a similar number of both non-smoking and tobacco smoking pregnant women for comparison. We will record a detailed record of e-cigarette and tobacco use by women during pregnancy as well as checking smoking using special monitoring tools. After the baby is born, we will perform growth measurements, neurocognitive assessments and a respiratory questionnaire at 6 months, one year and two years of age.

DETAILED DESCRIPTION:
Background Much is already known about the negative health effects of tobacco smoking during pregnancy. There is no national data on smoking in pregnancy but research indicates that up to 10% of Irish women continue to smoke tobacco in pregnancy. Tobacco smoking is associated with significant obstetric and perinatal complications including preterm birth, premature rupture of membranes, placental abruption, placenta previa and intrauterine growth restriction and stillbirth. Tobacco smoking is associated with a higher incidence of congenital abnormalities. Infants born to smoking mothers are at increased risk of necrotizing enterocolitis in the neonatal period, and of sudden infant death syndrome (SIDS). Children of smokers have an increased prevalence of wheeze and asthma. There is emerging evidence of cognitive impairment with higher rates of abnormal behavioural and neurodevelopmental outcomes such as attention deficit hyperactivity disorder (ADHD) and poor academic performance in the off-spring of mothers who smoke in pregnancy.

The popularity of electronic nicotine delivery systems (ENDS) has risen significantly over the past 10 years particularly among young adults and adolescents. ENDS (also called e-cigarettes or vaping devices) are battery powered devices that heat a solution (e-liquid) to create an aerosol that contains nicotine. In addition to nicotine, the e-liquid often contains different flavourings as well as the compounds Propylene Glycol and Glycerin. The vapour created by heating e-liquid at high temperatures alters the chemical profile of the original liquid by producing hazardous compounds such as aldehydes. More than 15,000 different flavours have been reported to date. ENDS aerosols contain fewer harmful substances when compared with tobacco smoking. As a result, they have been proposed as a safer alternative to tobacco smoking. Much research on these devices currently focuses on their role as a tobacco cessation tool. Currently there is insufficient evidence to determine if ENDS are a safe and effective long-term tobacco cessation method. However, there is emerging evidence that are not harmless products and that they contain toxic compounds which have hazardous effects on different organs in the body to users.

Research on the long-term health effects of ENDS, particularly from animal studies, suggests that there are negative growth, cardiopulmonary and neurological physiological changes caused by ENDS. Animal models have demonstrated that chronic exposure to ENDS results in increased arterial stiffness, vascular endothelial changes, increased angiogenesis and atherosclerotic plaque formation. Pulmonary changes including increased airway hyperreactivity, airway obstruction, inflammation and emphysematous changes have all been documented in animal studies on ENDS. Neurotoxic effects reported in mice studies include calcium dyshomeostasis, epigentic changes, impaired autophagy and neurotransmission, oxidate stress, mitochondrial dysfunction and neuroinflammation. As nicotine, the primary ingredient in ENDS, easily crosses the placental barrier; these harmful effects have the potential to impact the unborn foetus of pregnant women who use ENDS.

There is a paucity of real world data on the fetal and neonatal effects of ENDS use during pregnancy. A few studies which have examined obstetric and birth outcomes in women using e-cigarettes during pregnancy with mixed results. An Irish study of over 400 pregnant women reported that birth weight and neonatal outcomes were similar in women who were sole users of e-cigarettes when compared with non-smokers. However, two other studies did demonstrate an association between exclusive e-cigarette use during pregnancy and low birth weight and preterm delivery. These are important predictors of adverse outcomes in the neonatal period. The proposed study will help to clarify any association between ENDS use, preterm birth and fetal growth restriction.

The SNAP trial was a randomised control trial examining the effectiveness of nicotine replacement therapy (NRT) versus placebo on smoking cessation in pregnant women who smoked. The study also examined clinical outcomes at two years of age and found that children born to women on the NRT arm of the study had no adverse outcomes at two years of age. While NRT is generally considered a much safer option for pregnant women looking to quit smoking, ENDS are not currently recommended as a smoking cessation tool in Ireland or in most countries in the world. The use of ENDS among pregnant women has risen over the past decade. The exact prevalence of ENDS use is unknown but a number of studies across the world report this figure to be between 1-15%. A more recent systematic review from the US reported a prevalence of 1.2-7%, whereas the prevalence rate was 2.8% in a survey of over 4000 pregnant women in the UK.

According to the Healthy Ireland survey 2019, the current rate of ENDS use in Ireland is 5% and a further 12% have tried them at some point. Of those smokers who have made a quit attempt, 38% used ENDS. From an Irish perspective, we have very little data on the use of ENDS during pregnancy. A recent study from the Coombe Women & Infants University Hospital identified 449 pregnant ENDS over a period of 13 months (8500 deliveries per year). We expect that a similar number of ENDS users could be recruited at the other two Dublin maternity hospitals.

Knowledge gap At present, there is insufficient evidence on the clinical impact of prenatal exposure to ENDS on children. The hypotheses reported in animal studies need to be tested in longitudinal studies in humans. Real world studies are clearly needed to examine the impact of prenatal exposure of ENDS in childhood and beyond.

Research questions What are the nutritional, pulmonary, and neuro-behavioural consequences for young children born to mothers using ENDS during pregnancy?

The specific research questions are -

* Do infants exposed to ENDS in utero have a lower birthweight compared with infants of non-smokers?
* Are children exposed to ENDS in utero at a higher risk of wheeze/asthma at two years of age compared with children of non-smokers?
* Do children exposed to ENDS in utero have impaired neurocognitive functioning at the age of two years compared with children of non-smokers?
* Are these outcomes measures different between children exposed to ENDS in utero compared with children exposed to tobacco smoke in utero

Aims and objectives The aim of the ECHO study is to examine obstetric, growth, pulmonary, and neuro-behavioural outcomes over the first two years of life in children exposed to ENDS in utero and compare them with children born to pregnant women who are either tobacco smokers or non-smokers.

The objectives of the study are -

* To establish whether infants born to mothers who are ENDS users are at a higher risk of preterm birth compared with non-smokers but lower risk compared with smokers
* To establish whether there are significant differences in growth between children of women who use tobacco or ENDS and children of non-smokers
* To establish whether parent reported and doctor confirmed wheeze and/or asthma occurs more frequently in children exposed to ENDS in utero compared with children of non-smokers and less frequently compared with children of tobacco smokers
* To establish whether there are differences in healthcare utilisation between children exposed to tobacco smoking or ENDS in utero and children of non-smokers
* To establish whether there are significant differences in neurocognitive outcomes between children of women who use ENDS, women who smoke tobacco and children of non-smokers

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or greater and less than 46 years of age at booking
* Pregnant with a singleton fetus
* Smokers (exhaled CO reading of greater than or equal to 4) or
* Self-reported vaper or
* Dual user (smoker/vaper)
* Non-smokers
* Able to understand and read English.
* Willing to agree to follow-up for the two-year duration of the study in the postnatal period (ie. unlikely to move out of the catchment area).

Exclusion Criteria:

* Women pregnant with twins or higher order multiples
* Late bookers - defined as booking after 24+0 weeks' gestational age
* Fetus or infant diagnosed with a major congenital abnormality (major structural abnormality, ie congenital diaphragmatic hernia (CDH), omphalocele, major cardiac defects ie. which require immediate admission to NICU +/- transfer to cardiology for surgery, chromosomal abnormalities, syndromes - Turner's/Noonan's) or a lethal fetal anomaly
* Any inherited disorder of metabolism or Cystic Fibrosis on Guthrie Card/ neonatal blood spot screening
* History of significant medical disorder in pregnancy e.g. cardiac, haematological, or endocrine disease (including gestational diabetes requiring insulin)
* Significant maternal psychiatric disorder, e.g. delusional or psychotic disorders, severe depression requiring hospitalisation, use of >1 psychotropic drugs for treatment
* Serious co-morbid addiction issues e.g. opiate abuse, methadone maintenance program
* Severe intellectual disability or lack of capacity

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant woment
Study Population: The population under scrutiny in this prospective observational cohort are adult (18 to 46 years of age) women pregnant with a singleton, non-anomalous fetus, who can understand English and can give consent to partake in the study for its duration. Participants who smoke cigarettes, use vapes and controls will be invited to partake when they attend for the booking appointment at any of the Dublin maternity hospitals. They will be given written information about the study in their first visit booking back either in electronic or hardcopy format.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of preterm birth | Up to the time of birth
  Obstetric
Incidence of low birth weight | Up to the time of birth
  Neonatal: Defined as less than the 10th centile
Incidence of wheeze during the first two years of life | 6, 12 and 24 months
  Paediatric

SECONDARY OUTCOMES:
Incidence of smoking and vaping | Through study completion, up to 24 months
  Obstetric and paediatric
Estimated foetal weight | 20 and 34 weeks gestation
  Obstetric
Trends in carbon monoxide levels | Antenatal: At time of recruitment, 20 weeks, 34 weeks; postnatally: birth, 12 and 24 months
  Obstetric
Blood pressure measurements (both diastolic and systolic) | At time of recruitment, 20 weeks, 34 weeks
  Obstetric
Urine cotinine measurements | At time of recruitment, 20 weeks, 34 weeks and delivery
  Obstetric
Incidence of maternal cough, wheeze and/or asthma | At time of recruitment, 20 weeks, 34 weeks and birth
  Obstetric
Maternal history of abnormal cervical screening cytology | At time of recruitment
  Obstetric
Incidence of pre-eclampsia and/or hypertension during pregnancy | At time of recruitment, 20 weeks, 34 weeks and delivery
  Obstetric
Incidence of birth complications | At the time of birth
  Obstetric
Edinburgh postnatal depression score | At the time of birth
  Maternal neuropsychology (Scores are between 0 and 30, with scores 13 and above indicating depressive illness, or a high risk of developing a depressive disorder.)
APGAR scores at 1, 5 and 10 minutes after birth | At the time of birth
  Neonatal - APGAR: Appearance, Pulse, Grimace, Activity, Respiratory. Scores are between 0 and 10, with score above 7 normal.
Admission to neonatal intensive care | At the time of birth
  Neonatal
Incidence of neonatal complications | At the time of birth
  Neonatal
Neonatal and paediatric anthropometric measurements over first two years of life | At the time of birth, 12 and 24 months
  Neonatal and paediatric - (Weight, height, body mass index, head circumference, waist circumference, chest circumference and mid-arm circumference measurements)
Neonatal body composition measurements | At the time of birth
  Neonatal - using a PEA POD machine, we will measure measure body volume using air displacement plethysmography.
Incidence of respiratory illnesses | 6,12 and 24 months
  Paediatric
Number of attendances/admissions to hospital | 6,12 and 24 months
  Paediatric
Frequency of prescribed respiratory medications use | 6, 12 and 24 months
  Paediatric
Barkely Functional Impairment score (BFIS) | At the time of birth
  Maternal neuropsychology - The BFIS is designed to evaluate possible impairment in 15 major domains of psychosocial functioning in adults. The score is between 0-10, 10 being indicative of increased functional impairment.
Early Executive Functions Questionnaire (EEFQ) | 12 and 24 months
  Paediatric neuropsychology -The 31-item EEFQ parent report measure complements temperament measures by targeting cognitive and regulatory capabilities. Each question is scored between 1(never) and 7(always) to measure executive function in babies.
Infant Behaviour Questionnaire (IBQ) | 12 months
  Paediatric neuropsychology - The 37 item parent report measure of infant temperament. Each item is scored between 1 (never) and 7 (always to measure infant temperament.
Child Behaviour Checklist (CBCL) | 24 months
  Paediatric neuropsychology - The 113-item CBCL is a parent report measure designed to assess behavioural and emotional problems in children. The CBCL is scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often).
Early Childhood Behaviour Questionnaire (ECBQ) | 24 months
  Paediatric neuropsychology - The ECBQ is a parent reported measure of a child's temperament. The ECBQ contains 36 items with 7 broad likert scales from which a score is calculated. The higher the likert scale, the better the score.
Bayley Scales of Infant and Toddler Development (BSID) | 12 months
  Paediatric neuropsychology - The Bayley Scale is an extensive formal developmental assessment tool for diagnosing developmental delays in early childhood. The BSID measures scores in the five domains of cognition, language (receptive and expressive language abilities), motor skills (fine and gross motor skills), socio-emotional behaviour and adaptive behaviour. The BSID index scores within a range of 40-160. The higher score indicating normal development.

CONTACTS AND LOCATIONS:
Overall Officials: Des Cox, MB BCh BAO, Principal Investigator — University College Dublin
Locations (3):
- Ireland (3):
  - Rotunda Hospital, Dublin
  - National Maternity Hospital, Holles Street, Dublin
  - Coombe Womens Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

REFERENCES:
- [Background] Agarwal S, Trolice MP, Lindheim SR. E-cigarette use in reproductive-aged women and pregnancy: a rising health concern. Fertil Steril. 2020 Jun;113(6):1133-1134. doi: 10.1016/j.fertnstert.2020.01.031. Epub 2020 Mar 25. No abstract available. PMID 32222252
- [Background] Gould GS, Havard A, Lim LL, The Psanz Smoking In Pregnancy Expert Group, Kumar R. Exposure to Tobacco, Environmental Tobacco Smoke and Nicotine in Pregnancy: A Pragmatic Overview of Reviews of Maternal and Child Outcomes, Effectiveness of Interventions and Barriers and Facilitators to Quitting. Int J Environ Res Public Health. 2020 Mar 19;17(6):2034. doi: 10.3390/ijerph17062034. PMID 32204415
- [Background] Rogers JM. Tobacco and pregnancy. Reprod Toxicol. 2009 Sep;28(2):152-60. doi: 10.1016/j.reprotox.2009.03.012. Epub 2009 Apr 9. PMID 19450949
- [Background] Holbrook BD. The effects of nicotine on human fetal development. Birth Defects Res C Embryo Today. 2016 Jun;108(2):181-92. doi: 10.1002/bdrc.21128. Epub 2016 Jun 13. PMID 27297020
- [Background] Hsu G, Sun JY, Zhu SH. Evolution of Electronic Cigarette Brands From 2013-2014 to 2016-2017: Analysis of Brand Websites. J Med Internet Res. 2018 Mar 12;20(3):e80. doi: 10.2196/jmir.8550. PMID 29530840
- [Background] Ebell MH. e-Cigarettes More Effective Than Nicotine Replacement for Cessation of Tobacco Use in Adults. Am Fam Physician. 2019 Oct 1;100(7):442. No abstract available. PMID 31573159
- [Background] Hajek P, Phillips-Waller A, Przulj D, Pesola F, Myers Smith K, Bisal N, Li J, Parrott S, Sasieni P, Dawkins L, Ross L, Goniewicz M, Wu Q, McRobbie HJ. A Randomized Trial of E-Cigarettes versus Nicotine-Replacement Therapy. N Engl J Med. 2019 Feb 14;380(7):629-637. doi: 10.1056/NEJMoa1808779. Epub 2019 Jan 30. PMID 30699054
- [Background] Ibrahim S, Habiballah M, Sayed IE. Efficacy of Electronic Cigarettes for Smoking Cessation: A Systematic Review and Meta-Analysis. Am J Health Promot. 2021 Mar;35(3):442-455. doi: 10.1177/0890117120980289. Epub 2020 Dec 17. PMID 33327728
- [Background] Wang RJ, Bhadriraju S, Glantz SA. E-Cigarette Use and Adult Cigarette Smoking Cessation: A Meta-Analysis. Am J Public Health. 2021 Feb;111(2):230-246. doi: 10.2105/AJPH.2020.305999. Epub 2020 Dec 22. PMID 33351653
- [Background] Hartmann-Boyce J, McRobbie H, Lindson N, Bullen C, Begh R, Theodoulou A, Notley C, Rigotti NA, Turner T, Butler AR, Hajek P. Electronic cigarettes for smoking cessation. Cochrane Database Syst Rev. 2020 Oct 14;10(10):CD010216. doi: 10.1002/14651858.CD010216.pub4. PMID 33052602
- [Background] Tsai M, Byun MK, Shin J, Crotty Alexander LE. Effects of e-cigarettes and vaping devices on cardiac and pulmonary physiology. J Physiol. 2020 Nov;598(22):5039-5062. doi: 10.1113/JP279754. Epub 2020 Oct 12. PMID 32975834
- [Background] Gotts JE, Jordt SE, McConnell R, Tarran R. What are the respiratory effects of e-cigarettes? BMJ. 2019 Sep 30;366:l5275. doi: 10.1136/bmj.l5275. PMID 31570493
- [Background] Chun LF, Moazed F, Calfee CS, Matthay MA, Gotts JE. Pulmonary toxicity of e-cigarettes. Am J Physiol Lung Cell Mol Physiol. 2017 Aug 1;313(2):L193-L206. doi: 10.1152/ajplung.00071.2017. Epub 2017 May 18. PMID 28522559
- [Background] Ruszkiewicz JA, Zhang Z, Goncalves FM, Tizabi Y, Zelikoff JT, Aschner M. Neurotoxicity of e-cigarettes. Food Chem Toxicol. 2020 Apr;138:111245. doi: 10.1016/j.fct.2020.111245. Epub 2020 Mar 5. PMID 32145355
- [Background] Breland A, McCubbin A, Ashford K. Electronic nicotine delivery systems and pregnancy: Recent research on perceptions, cessation, and toxicant delivery. Birth Defects Res. 2019 Oct 15;111(17):1284-1293. doi: 10.1002/bdr2.1561. Epub 2019 Jul 31. PMID 31364280
- [Background] Greene RM, Pisano MM. Developmental toxicity of e-cigarette aerosols. Birth Defects Res. 2019 Oct 15;111(17):1294-1301. doi: 10.1002/bdr2.1571. Epub 2019 Aug 9. PMID 31400084
- [Background] McDonnell BP, Dicker P, Regan CL. Electronic cigarettes and obstetric outcomes: a prospective observational study. BJOG. 2020 May;127(6):750-756. doi: 10.1111/1471-0528.16110. Epub 2020 Feb 9. PMID 32036628
- [Background] Wang X, Lee NL, Burstyn I. Smoking and use of electronic cigarettes (vaping) in relation to preterm birth and small-for-gestational-age in a 2016 U.S. national sample. Prev Med. 2020 May;134:106041. doi: 10.1016/j.ypmed.2020.106041. Epub 2020 Feb 24. PMID 32105682
- [Background] Kim S, Oancea SC. Electronic cigarettes may not be a "safer alternative" of conventional cigarettes during pregnancy: evidence from the nationally representative PRAMS data. BMC Pregnancy Childbirth. 2020 Sep 23;20(1):557. doi: 10.1186/s12884-020-03247-6. PMID 32967660
- [Background] Cooper S, Lewis S, Thornton JG, Marlow N, Watts K, Britton J, Grainge MJ, Taggar J, Essex H, Parrott S, Dickinson A, Whitemore R, Coleman T; Smoking, Nicotine and Pregnancy Trial Team. The SNAP trial: a randomised placebo-controlled trial of nicotine replacement therapy in pregnancy--clinical effectiveness and safety until 2 years after delivery, with economic evaluation. Health Technol Assess. 2014 Aug;18(54):1-128. doi: 10.3310/hta18540. PMID 25158081
- [Background] Cooper S, Taggar J, Lewis S, Marlow N, Dickinson A, Whitemore R, Coleman T; Smoking, Nicotine and Pregnancy (SNAP) Trial Team. Effect of nicotine patches in pregnancy on infant and maternal outcomes at 2 years: follow-up from the randomised, double-blind, placebo-controlled SNAP trial. Lancet Respir Med. 2014 Sep;2(9):728-37. doi: 10.1016/S2213-2600(14)70157-2. Epub 2014 Aug 10. PMID 25127405
- [Background] Kapaya M, D'Angelo DV, Tong VT, England L, Ruffo N, Cox S, Warner L, Bombard J, Guthrie T, Lampkins A, King BA. Use of Electronic Vapor Products Before, During, and After Pregnancy Among Women with a Recent Live Birth - Oklahoma and Texas, 2015. MMWR Morb Mortal Wkly Rep. 2019 Mar 1;68(8):189-194. doi: 10.15585/mmwr.mm6808a1. PMID 30817748
- [Background] Cardenas VM, Fischbach LA, Chowdhury P. The use of electronic nicotine delivery systems during pregnancy and the reproductive outcomes: A systematic review of the literature. Tob Induc Dis. 2019 Jul 1;17:52. doi: 10.18332/tid/104724. eCollection 2019. PMID 31582941
- [Background] Opondo C, Harrison S, Alderdice F, Carson C, Quigley MA. Electronic cigarette use (vaping) and patterns of tobacco cigarette smoking in pregnancy-evidence from a population-based maternity survey in England. PLoS One. 2021 Jun 4;16(6):e0252817. doi: 10.1371/journal.pone.0252817. eCollection 2021. PMID 34086809
- [Derived] Healy EF, O'Connell A, Yousef MS, Reddin A, Boyle M, Coleman T, Doolan A, Fitzpatrick P, Frazer K, Higgins S, Kelleher C, Malone FD, O'Currain E, Seguardo R, Walsh J, Cox D, Downes M, Regan C. The impact of electronic cigarettes on pregnancy and childhood health outcomes: the ECHO study-a protocol for a multicentre, prospective, observational, cohort. Arch Gynecol Obstet. 2025 Sep;312(3):927-935. doi: 10.1007/s00404-025-08066-8. Epub 2025 Jun 20. PMID 40540019